CLINICAL TRIAL: NCT02211287
Title: Promoting Informed Decision Making and Effective Communication Through Advance Care Planning for People With Dementia and Their Family Carers
Brief Title: Promoting Informed Decision Making Through Advance Care Planning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queen's University, Belfast (Other)
Collaborators: Four Seasons Health Care (Unknown)
Responsible Party: Principal Investigator, Kevin Brazil, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: B14/25
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-04

CONDITIONS: Dementia; Neurodegenerative Diseases
Keywords: Dementia; Decision-making; Communication; Advance Care Planning
MeSH Terms: conditions — Dementia; Neurodegenerative Diseases; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention will include five key elements: a Project Nurse - ACP facilitator; family education on comfort care at the end of life for individuals with dementia using the 'Comfort Care at the end of life for persons with dementia' booklet; a family meeting with follow-up telephone call; documentation of ACP decisions, and orientation and education directed towards General Practitioners (GPs) and nursing home staff about the intervention.
  Interventions: Other: 'Comfort Care at the End of Life for Persons with Dementia'; Other: Project Nurse - ACP Facilitator
- Usual care (No Intervention): Care will continue as usual for the nursing home residents

INTERVENTIONS:
Other: 'Comfort Care at the End of Life for Persons with Dementia' — A guide for caregivers to provide information on the trajectory of the disease, clinical issues, decision-making processes, and symptom management. The guide is written in a Q&A form and can help answer frequent family questions.
  Arms: Intervention
Other: Project Nurse - ACP Facilitator — A nurse will receive training in the 'Respecting Choices Facilitator Curriculum' - an online program consisting of a series of six critical thinking modules designed for healthcare professionals who want to enhance their ACP facilitation skills. Local training resources in Northern Ireland will supplement.
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate the application of a best-practice Advance Care Planning (ACP) model for individuals living with dementia in a sample of nursing homes in Northern Ireland

ELIGIBILITY:
Inclusion Criteria:

1. Family Caregivers

   * Family caregivers of a resident who does not have decision making capacity to participate in ACP discussion
   * Individuals identified by the nursing home manager as the family member who possess power of attorney for personal care and/or viewed by the nursing home staff as most involved in the care of the resident who does not have decision making capacity.
2. Health Care Professionals

Nursing home managers, registered nursing staff and GPs who:

* are employed, or in the case of GPs, care for residents, in the six nursing homes that were part of the intervention group
* were familiar with the intervention to discuss its strengths and weaknesses in an interview
* are able to speak English as they are required to participate in interviews.

Exclusion Criteria:

* Family caregivers and health care professionals who are unable to communicate through written and spoken English.
* Family caregivers who has a family resident considered to have the ability to participate in ACP discussions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Primary Completion 2015-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Level of family carer satisfaction in decision making about the care of the resident | Baseline, up to 2 months
  Decisional Conflict Scale (DCS). This measures uncertainty and difficulties in the decision making process. The 16 item version measures four domains: a) uncertainty in choosing options; b) unsupported in decision making; c) feeling informed; d) decision is consistent with values

SECONDARY OUTCOMES:
The level of family carer satisfaction with nursing home care | Baseline up to 2 months
  The Family Perception of Care Scale (FPCS). This instrument will represent a global measure on the quality of nursing home care. It is comprised of four subscales: 1) resident care, 2) family support, 3) communication, and 4) rooming. One can investigate both the total and the subscale scores. Family members will also be asked to identify three of the 25 items in the instrument as the highest priorities for providing quality care in the nursing home. Respondents will also be invited to include written comments.
Level of family carer anxiety and depression | Baseline up to 2 months
  General Health Questionnaire (GHQ-12). This 12-item instrument is a self-report measure of psychological morbidity. It is widely used in clinical practice, epidemiological research and for research in psychology. The GHQ-12 is often used to assess general distress. It is designed to cover four identifiable elements of distress: anxiety, depression, social impairment, and hypochondriasis.
The comfort of the resident at the end of life | Baseline up to 2 months
  Quality of Dying in Long Term Care (QoDLTC). This instrument is a retrospective scale representing psychosocial aspects of quality of dying. The questionnaire contains 11 items with three subscales: personhood (5 items), closure (3 items) and preparatory tasks (3 items). Factor scores (means of item scores within each factor) may be averaged for an overall quality of dying score (range 1 - 5), with a higher score indicating a more positive experience. Individual factor scores may also be used separately.
Number of unnecessary hospitalisations | Baseline up to 12 months
  Assessed through the facility care home administrative records

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Brazil, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Four Seasons Health Care -- Nursing Homes, Belfast, United Kingdom